CLINICAL TRIAL: NCT04637360
Title: To Study the Bone Turnover Markers and Bone Density Changes in Hyperperparathyroid Dialysis Patients Under Calcium Sensing Receptor Agonist Cinacalcet Treatment
Brief Title: Bone Markers and Bone Density Changes in Hyperperparathyroid Dialysis Patients Under Cinacalcet Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Min-Sheng General Hospital (Other)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other); Taipei Medical University (Other); En Chu Kong Hospital (Other); National Taiwan University (Other); Taichung Tzu Chi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSIRB2018004
Record Dates: First submitted 2020-11-06; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Hyperparathyroidism; Secondary, Renal
Keywords: clastokines; hemodialysis; hyperparathyroidism; osteoporosis
MeSH Terms: conditions — Hyperparathyroidism; Neoplasm Metastasis; Osteoporosis | interventions — Cinacalcet; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinacalcet treatment (Experimental): hyperparathyroid dialysis patients using cinacalcet and active vitamin D for 6 months
  Interventions: Drug: Cinacalcet Tablets; Drug: calcitriol
- traditional therapy active vitamin D (Experimental): hyperparathyroid dialysis patients using traditional therapy active vitamin D without use cinacalcet for 6 months.
  Interventions: Drug: calcitriol

INTERVENTIONS:
Drug: Cinacalcet Tablets — All study subjects were treated with a fixed dose of oral Cinacalcet (25 mg/day) from baseline to 6 months.
  Other Names: CINACA®, Anxo, Taiwan
  Arms: Cinacalcet treatment
Drug: calcitriol — All hyperparathyroidism were treated as traditional therapy with oral calcitriol 0.25 mcg(dosage according to IPTH serum level) from baseline to 6 months.
  Other Names: Macalol Cap 0.25mcg

SUMMARY:
Chronic kidney disease related mineral and bone disorders (CKD-MBDs) and secondary hyperparathyroidism (SHPT) are observed in most patients with chronic kidney disease on dialysis (CKD-5D). The original use of the calcimimetic cinacalcet in these patients was to reduce the elevated parathyroid hormone (PTH) levels; however, subsequent clinical studies consistently confirmed its beneficial effects on mineral disturbances and bone disease. Although many mechanisms proposed, its specific mechanisms underlying the bone disease is still unclear. Recently, Wnt signaling and their inhibitors were proposed to involve in fine control of osteoclast-to-osteoblast cross-talk. In previous study, investigators explore the changes in Wnt 10b in bone microenvironment after addition of calcimimetic cinacalcet using in vitro osteoclasts. In vitro results were confirmed in 5/6 nephrectomy mice, which were grouped into control, with cinacalcet and without cinacalcet groups. From in-vitro study, investigators found cinacalcet increase mineralization; enhance osteoclast apoptosis, which probably work as osteoclast-osteoblast cross talk for bone formation. Similar results were found in-vivo animal study, and the micro-CT of cinacalcet treated CKD animals revealed a significantly decrease in cortical porosity. On the basis of our in-vitro and animal study, investigators propose that cinacalcet have definitive role on bone turnover marker and bone density changes among SHPT dialysis patients.

Methods: Our study includes 50 hyperparathyroid dialysis patients using cinacalcet from 1st Dec 2017 to 31 Oct 2018. Investigators will exclude post-menopausal female subjects. Enzyme-linked immunosorbent assay and Western blot analysis will be done for bone turnover markers (TRACP，Alk-P，S1P，BMP6，Wnt，10B，16，SOST，P1NP，PDGF BB，HGF and CTHRC1, etc.). Bone mineral density will be determined by dual-energy X-ray absorptiometry (DXA). Plasma fibroblast growth factor (FGF-23), Ca 2+ , P 3+ , calcium-phosphorus product and parathyroid hormone will also be measured. Data will be collected and analyzed the differences between baseline measures and 4 weekly and follow up for 6 months after the treatment. Control group that we enrolled 30 hyperparathyroid dialysis patients using traditional therapy active vitamin D without use cinacalcet.

DETAILED DESCRIPTION:
BACKGROUND Secondary hyperparathyroidism (SHPT) is an important mechanism underlying most cardiovascular and bone turnover disorders in CKD-5D patients, which contribute highest morbidity and mortality annually. Impair phosphate excretion and failure to bioactivate vitamin D during progressive renal function deterioration continuously stimulates the synthesis and secretion of parathyroid glands. Increase serum phosphate stimulates the phosphatonin fibroblast growth factor 23 (FGF-23) releases from osteocytes and osteoblasts. Elevated FGF-23 downregulates renal 25(OH)-1-hydroxylase which further deteriorates SHPT. Prolonged parathyroid gland functional activation leads to progressive parathyroid hyperplasia. Downregulation of the parathyroid vitamin D receptors and calcium-sensing receptors occurs within parathyroid gland, and principally responsible for the parathyroid hyperplasia. Hyperparathyroidism and alteration in mineral metabolism, especially hyperphosphatemia, modulate renal osteodystrophy and vascular calcification (together known as CKD-MBD). Continuously high PTH during SHPT stimulates osteoclastic resorption and bone remodeling rates, which leads to classic osteitis fibrosa. Excessive osteoblast viability and activity because of persistent hyperparathyroidism may follow to compensate for the bone resorption, with resultant osteosclerosis. Metastatic calcification and vascular calcification occur as a result of increased calcium and phosphate solubility product in extracellular fluid. The degree of mineralization is impaired in those with a high-turnover status because the recently formed bone is removed rapidly without adequate mineralization. Bones from a high-turnover state have lower mineralization and lower trabecular microhardness than do bones from normal or low-turnover states. A low mineral-to-matrix ratio and low carbonate-to-phosphate ratio reduce bone toughness. Moreover, collagen crosslinking abnormalities have been observed in both serum and soft tissue, which were responsible for bone quality in these patients. High PTH also generates microstructural damage at both the cortical and trabecular levels in CKD patients. Specifically, with chronic excess PTH secretion, increased catabolism and decreased cortical thickness is noted in cortical bone; whereas in trabecular bone, increased trabecular thickness with disturbed trabecular quality are noted. Taking together, SHPT patients have a higher risk of skeletal fractures and poor clinical outcomes associated with both bone quantity and quality loss.

Clinically, bone histomorphometry is still considered as the gold standard though clinically unfeasible due to its invasive and technician-dependent nature. Serum intact PTH (iPTH) and BSAP are recently used as markers of turnover to discriminate renal osteodystrophy. High serum iPTH and BSAP considered as high-turnover bone disease, whereas low serum iPTH, low BSAP, and normal vitamin D levels occur in adynamic bone disease (ABD) patients. Low vitamin D and PTH levels in conjunction with high levels of BSAP are correlated with osteomalacia. The Kidney Disease Outcomes Quality Initiative (K/DOQI) guideline use intact parathyroid hormone (iPTH) as a reliable surrogate marker for bone turnover and suggested that iPTH should be maintained in a target range between 150 and 300 pg ml-1 for patients with stage 5 CKD patients. However, some studies33 also found discrepancies between iPTH and histomorphometry findings in dialysis patients. Bone-derived markers of bone formation and resorption may be required to accurately measure bone structure and function in these patients. Bone formation markers including bone-specific alkaline phosphatase (BSAP), osteocalcin, and procollagen type-1 N-terminal propeptide (P1NP) are markers of osteoblast function. Bone resorption markers such as tartrate-resistant acid phosphatase 5b (Trap-5b) and C-terminal telopeptides of type I collagen (CTX) are markers of osteoclast number and function. Trap-5b and BSAP are not cleared by the kidneys and are mostly used in CKD patients as useful biomarkers. Osteocalcin, P1NP monomer, and CTX are cleared by the kidneys, and their usefulness in treating CKD patients remains unclear. Although many other circulating markers for bone remodeling disorders in CKD 34 patients have been evaluated, their clinical uses still not clear.

Human genetic studies have highlighted the crucial role of wingless (Wnt) signaling in bone mass regulation. Wnts are extracellular proteins that are linked to intracellular canonical and noncanonical Wnt signaling pathways when activated. They were found to be implicated in osteoblast and osteoclastic differentiation and function35, which are critical for trabecular and cortical bone mass. Wnt3a and Wnt10b, acting through canonical signaling; and Wnt16, acting through both canonical and noncanonical signaling, induce production of OPG in osteoblasts. OPG binds to the osteoclast-inducing cytokine RANKL and thereby inhibits osteoclast differentiation. Osteoblast Wnt5a potentiates RANK-induced osteoclast differentiation by activating ROR2-dependent noncanonical signaling. By contrast, Wnt 4 and Wnt 16 act directly through noncanonical signaling on osteoclast progenitors to inhibit RANKL-induced osteoclast formation. In addition to these known concepts about osteoblast-lineage cells influence on osteoclast precursors, recent researchers found that osteoclasts are capable of producing 'clastokines' that regulate osteoblast performance and bone formation. A study demonstrated that osteoclasts recruit osteoprogenitors and promote mineralization through the release of chemokine sphingosine 1 phosphate(S1P), bone morphogenetic protein 6 (BMP6) and Wnt10b. Further, osteoclast production of Wnt 10b found to mediate mineralization through increased TGF-βduring bone resorption phase. The sophisticated role of Wnt signaling in the human CKD and end-stage renal disease (ESRD) population still requires exploration. Several therapeutic interventions (active vitamin D analogues, phosphate binders, calcimimetics or surgical parathyroidectomy) are used nowadays to modulate mineral disturbances in order to reduce the CKD-MBD related clinical consequences. Calcimimetics, such as cinacalcet, a positive allosteric modulator of the calcium sensing receptor (CaSR), increases the PTH sensitivity to extracellular calcium and subsequently reduces the PTH secretion. Extensive preclinical studies have indicated that calcimimetics also arrest the progression of parathyroid hyperplasia. Combined randomized clinical trials (RCTs) and phase 4 studies confirmed the pleiotropic effects of calcimimetic agents in clinical grounds, including reduction of the elevated bone formation rate/tissue area with improvement in high turnover bone disorders. Some studies also confirm that adding calcimimetic cinacalcet can reduce the risk of fractures in SHPT patients. A bone histomorphologic study of 4 HD patients under cinacalcet treatment revealed decreased bone fibrosis, osteoblast surface and osteoid-related parameters.

Although mechanisms of calcimimetics in parathyroid hyperplasia are clearly explored, its effects on osteoclasts and osteoblasts (basic multicellular units) at bone remodeling sites are still unclear. A study revealed high extracellular calcium induces mitogenic action of osteoblasts via calcium-sensing receptors. However, another in vitro study on mouse and human adult osteoclastic and osteoblastic cells demonstrated the calcium dependent increase osteoblast formation and decrease osteoclast formation/function might not through the calcium sensing receptors, and not effected by calcimimetics. The calcimimetics might have any other mechanisms not through effects on calcium or calcium sensing receptors on these osteoblasts. Based on above information, investigators hypothesized that bone turnover markers including Wnt changes occur in SHPT hemodialysis patients. In addition, investigators consider the hypothetical role of cinacalcet mediated bone turnover changes occurred in the process of cinacalcet related bone anabolism.

ELIGIBILITY:
Inclusion Criteria:

1. 20 - 80 yrs of age and eligible for consent
2. Hyperparathyroid (iPTH>300 pg/mL) regular dialysis patients using cinacalcet and start the treatment during the study period.

Exclusion Criteria:

1. <20yrs or >80yrs patients
2. Post-menopausal female patients
3. Malignancies, inflammatory or infectious disease < 3 months
4. Pregnancy
5. Severe malnutrition
6. Surgical intervention < 3 months
7. Acute myocardial infarction, unstable angina, cerebrovascular disease or transient ischemic attack, deep vein thrombosis, pulmonary embolism, congestive heart failure < 3months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Parathyroid serum level | After treatment for 6 months.
  lower in serum intact parathyroid serum level (iPTH<300 pg/mL) with 6 months cinacalcet treatment.

SECONDARY OUTCOMES:
Bone mineral density | After treatment for 6 months.
  Improve bone mineral density (dual-energy x-ray absorptiometry (DXA)) with 6 months cinacalcet treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ren-Si Syu, Dr., Study Director — Min-Sheng General Hospital
Locations (1):
- Min sheng general hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Work Group. KDIGO clinical practice guideline for the diagnosis, evaluation, prevention, and treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl. 2009 Aug;(113):S1-130. doi: 10.1038/ki.2009.188. PMID 19644521
- [Background] London GM, Marchais SJ, Guerin AP, Boutouyrie P, Metivier F, de Vernejoul MC. Association of bone activity, calcium load, aortic stiffness, and calcifications in ESRD. J Am Soc Nephrol. 2008 Sep;19(9):1827-35. doi: 10.1681/ASN.2007050622. Epub 2008 May 14. PMID 18480316
- [Background] Cunningham J, Locatelli F, Rodriguez M. Secondary hyperparathyroidism: pathogenesis, disease progression, and therapeutic options. Clin J Am Soc Nephrol. 2011 Apr;6(4):913-21. doi: 10.2215/CJN.06040710. Epub 2011 Mar 31. PMID 21454719
- [Background] Westin G, Bjorklund P, Akerstrom G. Molecular genetics of parathyroid disease. World J Surg. 2009 Nov;33(11):2224-33. doi: 10.1007/s00268-009-0022-6. PMID 19373510
- [Background] Zheng CM, Zheng JQ, Wu CC, Lu CL, Shyu JF, Yung-Ho H, Wu MY, Chiu IJ, Wang YH, Lin YF, Lu KC. Bone loss in chronic kidney disease: Quantity or quality? Bone. 2016 Jun;87:57-70. doi: 10.1016/j.bone.2016.03.017. Epub 2016 Apr 2. PMID 27049042
- [Result] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Result] Mazzaferro S, Tartaglione L, Rotondi S, Bover J, Goldsmith D, Pasquali M. News on biomarkers in CKD-MBD. Semin Nephrol. 2014 Nov;34(6):598-611. doi: 10.1016/j.semnephrol.2014.09.006. PMID 25498379